CLINICAL TRIAL: NCT05338892
Title: Outcomes in Patients With Relapse/Refractory Diffuse Large B-Cell Lymphoma Treated With Systemic Therapy From Real-World Experience (ORCHID)
Brief Title: Real-World Clinical Outcomes in Adult Patients Who Initiate Systemic Treatment for Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Acronym: ORCHID
Status: Completed | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R1979-ONC-2090
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: Relapsed/Refractory Diffuse Large B-Cell Lymphoma (r/r DLBCL); Non-Hodgkin lymphoma; Chronic lymphocytic leukemia; Follicular lymphoma; Odronextamab; ORCHID
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with r/r DLBCL who were treated with at least 2 prior systemic therapies in the real-world setting
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — No study treatment will be administered on this study.

SUMMARY:
Primary Objective:

To evaluate objective response rate (ORR) in adult patients with Relapsed/Refractory Diffuse Large B-Cell Lymphoma (r/r DLBCL) who receive systemic treatment after at least 2 prior systemic therapies in the real-world setting according to Lugano classification of malignant lymphoma (Cheson, 2014) and as assessed by independent central review

Secondary Objectives:

To evaluate the following outcomes in adult patients with r/r DLBCL who are treated with currently available therapies in the real-world setting:

1. ORR according to Lugano classification and as assessed by treating physician evaluation
2. Complete Response (CR) rate according to Lugano classification and as assessed by:

   * Independent central review, and
   * Treating physician evaluation
3. Progression Free Survival (PFS) according to Lugano classification and as assessed by:

   * Independent central review, and
   * Treating physician evaluation
4. Overall Survival (OS)
5. Duration of response (DOR) according to Lugano classification and as assessed by

   * Independent central review and
   * Treating physician evaluation
6. Disease control rate (DCR) according to Lugano classification and as assessed by:

   * Independent central reviewed
   * Treating physician evaluation
7. Time to next treatment (TTNT)

ELIGIBILITY:
Key Inclusion Criteria:

1. Have a histologically confirmed diagnosis of DLBCL on or after 01 Jan 2010 as defined in the protocol
2. Have been r/r to at least 2 lines of systemic therapy for DLBCL, including an anti-CD20 antibody and an alkylating agent as defined in the protocol
3. Have initiated at least one additional line (3L+) of systemic therapy (salvage therapy) for DLBCL between 01 Jan 2015 and 30 Jun 2021 (indexing period) after meeting the criteria for r/r DLBCL as described above; the first additional line of systemic therapy during the indexing period that meets all of the remaining inclusion and exclusion criteria defined below will be the patients' first qualifying salvage therapy.
4. Have measurable disease on cross sectional imaging (defined as at least 1 bi-dimensionally measurable nodal lesion ≥1.5 centimeter [cm] in the greatest transverse diameter [GTD] regardless of the short axis diameter) documented by diagnostic imaging (computed tomography [CT], or magnetic resonance imaging [MRI]) recorded on or during the 8 weeks prior to index date
5. Have been seen at a site that routinely assesses DLBCL treatment response according to Lugano classification of malignant lymphoma (ie, sites with ≥50% DLBCL patients with treatment response according to Lugano classification)
6. Have DLBCL treatment response assessed according to Lugano classification of malignant lymphoma or are deceased prior to opportunity for assessment

Key Exclusion Criteria:

1. Primary central nervous system (CNS) lymphoma or known involvement by non-primary CNS non-Hodgkin's lymphoma (NHL) on or prior to index date
2. History of allo-stem cell transplant (SCT) prior to index date
3. Treatment with any chimeric antigen receptor T (CAR-T) therapy prior to index date
4. Received anti-CD20 x anti-CD3 bispecific therapy prior to index date
5. History of neurodegenerative condition or CNS movement disorder on or prior to index date
6. Evidence of significant cardiovascular disease on or prior to index date
7. Evidence of significant pulmonary disease, defined as obstructive pulmonary disease and a history of symptomatic bronchospasm on or prior to index date
8. Eastern Cooperative Oncology Group (ECOG) performance status >1 on or prior to index date
9. Inadequate organ function as defined in the protocol

Note: Other protocol-defined Inclusion/Exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with DLBCL who have relapsed after or are refractory to at least 2 prior lines of systemic therapy, including an anti-CD20 antibody and an alkylating agent.
Sampling Method: Probability Sample
Enrollment: 595 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Up to 84 months
  The proportion of best overall response of complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Complete Response (CR) rate | Up to 84 months
  The proportion of patients with a CR after initiation of the selected line of therapy (LoT).
Progression Free Survival (PFS) | Up to 84 months
  The time from the start date of the selected LoT until the first date of progressive disease (PD) or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to 84 months
  The time from the start date of the selected LoT until death due to any cause.
Duration of Response (DOR) | Up to 84 months
  The time from the date of the first documented CR or PR until the first date of PD or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | Up to 84 months
  The proportion of patients who achieve a best overall response of CR, PR, or stable disease (SD).
Time to Next Treatment (TTNT) | Up to 84 months
  The time from the start date of the selected LoT to the start of a new antineoplastic treatment line.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (9):
- Regeneron Research Facility, Graz, Austria
- France (3):
  - Regeneron Research Facility, Caen
  - Regeneron Research Facility, Paris
  - Regeneron Research Facility, Pierre-Bénite
- Germany (2):
  - Regeneron Research Facility, Essen
  - Regeneron Research Facility, Frankfurt
- United Kingdom (3):
  - Regeneron Research Facility, London
  - Regeneron Research Facility, Manchester
  - Regeneron Research Facility, Nottingham

IPD SHARING:
Plan to Share IPD: No